CLINICAL TRIAL: NCT04514796
Title: A Randomised, Single-blind, Two-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity of Two Formulations of SB5 in Healthy Male Subjects
Brief Title: Pharmacokinetics, Safety, Tolerability, and Immunogenicity of Two Formulations of SB5 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SB5-1003
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Healthy
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 40 mg/0.4 mL of SB5 (Experimental): 100 mg/mL of SB5
  Interventions: Drug: Adalimumab
- 40 mg/0.8 mL of SB5 (Active Comparator): 50 mg/mL of SB5
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — SB5 (adalimumab), 40 mg, single-dose

SUMMARY:
This study is to evaluate to compare the pharmacokinetics, safety, tolerability, and immunogenicity of two formulations of SB5 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria

1. Healthy male, aged 18-55 years (inclusive).
2. A body weight between 65.0-90.0 kg (inclusive) and a body mass index between 20.0-29.9 kg/m2 (inclusive)
3. 12-lead electrocardiogram results without clinically significant abnormal.
4. Systolic blood pressure ≤ 140 and ≥ 90 mmHg, diastolic blood pressure ≤ 90 and ≥ 50 mmHg and pulse rate ≥ 45 and ≤ 90 beats per minute or assessed as not clinically significant.
5. Physical examination results without clinically significant abnormal findings.
6. Clinical laboratory results within the normal range or outside the normal range but assessed as not clinically significant.
7. Male subjects who did not have surgical sterilisation must be willing to abstain from sexual intercourse or willing to use a condom in addition to having their female partner use another form of contraception such as an intra-uterine device, oral contraceptive, injectable progesterone, sub-dermal implant, or a tubal ligation unless their partners are infertile from the time of the investigational product (IP) administration until 5 months after the IP administration.
8. Willing and able to comply with study procedures including lifestyle consideration.
9. Able to provide written informed consent prior to any study procedures.

Exclusion Criteria

1. A history and/or current presence of clinically significant atopic, hypersensitivity or allergic, also including known or suspected clinically relevant drug hypersensitivity to adalimumab or to any of the excipients.
2. A history of and/or current clinically significant gastrointestinal, renal, hepatic, haematological, pulmonary, neurologic, psychiatric, drug or alcohol abuse, or allergic disease excluding mild asymptotic seasonal allergies.
3. Either active or latent tuberculosis (TB) or a history of TB.
4. A history of invasive systemic fungal infections or other opportunistic infections.
5. A history of any systemic or local infection, a known risk for developing sepsis and/or known active inflammatory process within 180 days prior to Randomisation.
6. A sign of ongoing or chronic inflammation process defined as high blood concentration of C reactive protein (> 1.5 times the upper limit of normal).
7. A history of serious infection (associated with hospitalisation and/or which required intravenous antibiotics) within 180 days prior to Randomisation.
8. Previously been treated with adalimumab.
9. Previously been exposed to a monoclonal antibody or fusion protein (other than adalimumab) within 180 days prior to Randomisation and/or there is a confirmed evidence or clinical suspicion of immunogenicity from previous exposure to a monoclonal antibody or fusion protein.
10. Previously been exposed to an immunosuppressive agent or biological agent (any other than a monoclonal antibody or fusion protein) within 120 days prior to Randomisation.
11. Received live vaccine(s) within 30 days prior to Randomisation or who will require live vaccine(s) during the study period.
12. A history of and/or current cardiac disease defined as one of the following:

    1. Personal or family history of prolonged QT interval syndrome or Torsade de Pointes.
    2. QT interval corrected by Fridericia's formulas > 450 msec or PR interval outside the range 120 to 220 msec.
    3. Signs and symptoms or any history suggestive for heart failure.
    4. Any other cardiac abnormalities or conditions assessed as clinically significant.
13. Impaired liver, pancreas and biliary system as determined by one of the following:

    1. Serum alanine transaminase and/or aspartate transaminase ≥ 1.5 times the upper limit of normal.
    2. Gallbladder or bile duct disease classified as clinically significant.
    3. Acute or chronic pancreatitis.
    4. A positive hepatitis C virus antibody test or hepatitis B virus surface antigen test, or signs for active or chronic hepatitis B.
    5. Hepatic disease classified as clinically significant.
14. A positive test result for human immunodeficiency virus, or have a history of immunodeficiency.
15. A history of malignancy (including lymphoma and leukaemia) other than a successfully treated non-metastatic cutaneous squamous cell carcinoma, basal cell carcinoma or localised carcinoma.
16. Had surgery within 90 days prior to Randomisation, and/or who plan to have an operation during the study period.
17. A history and/or current presence of an illness within 14 days prior to Randomisation that is classified as clinically significant.
18. Have a history of and/or current Coronavirus Disease-19 (COVID-19) defined as one of the following:

    1. Positive test result for COVID-19 confirmed by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) using real-time reverse transcriptase polymerase chain reaction (RT-PCR) at Day -1.
    2. Signs and symptoms consistent with COVID-19 30 days prior to Randomisation.
    3. Have had a positive test result for COVID-19 confirmed by SARS-CoV-2 detection using real-time RT-PCR.
    4. Had severe course of COVID-19.
19. Smoked more than 10 cigarettes, 2 cigars or 2 pipes per day within 90 days prior to Screening.
20. Regular consumption of alcoholic beverages that exceeds 14 units.
21. A positive urinary drug screening result.
22. Any prescription medicine or over-the-counter medicines (except paracetamol) that might have an effect on the objectives of the study in the opinion of the Investigator, within 30 days prior to Randomisation.
23. Donated > 100 mL blood or plasma within 28 days prior to Randomisation.
24. Participated in another study with an investigational drug within 60 days prior to Randomisation or are currently participating in or intending to participate in another clinical study of an investigational drug before completion of all scheduled evaluations in this clinical study.
25. Subjects who, in the opinion of the Investigator, are not likely to complete the study for whatever reason.
26. Subject who is the Investigator or any sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the clinical study.
27. Vulnerable subjects.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
AUCinf | Day 1 to Day 57
  Area under the concentration-time curve from time zero to infinity
Cmax | Day 1 to Day 57
  Maximum serum concentration

SECONDARY OUTCOMES:
AUClast | Day 1 to Day 57
  Area under the concentration-time curve from time zero to the last quantifiable concentration
Tmax | Day 1 to Day 57
  Time to reach Cmax
Vz/F | Day 1 to Day 57
  Apparent volume of distribution during the terminal phase
λz | Day 1 to Day 57
  Terminal rate constant
t1/2 | Day 1 to Day 57
  Terminal half-life
CL/F | Day 1 to Day 57
  Apparent total body clearance
%AUCextrap | Day 1 to Day 57
  Percentage of AUCinf due to extrapolation from time of last measurable concentration (Tlast) to infinity
Incidence of treatment-emergent adverse events (TEAEs) | Day 1 to Day 57
  Experience at least 1 TEAE
Incidence of serious adverse events (SAEs) | Day 1 to Day 57
  Experience at least 1 SAE
Incidence of anti-drug antibodies (ADAs) | Day 1 to Day 57
  Incidence of ADAs to adalimumab
Incidence of neutralising antibodies (NAbs) | Day 1 to Day 57
  Incidence of NAbs to adalimumab

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Köernicke, MD, Principal Investigator — Parexel International GmbH, Early Phase Clinical Unit Berlin
Locations (1):
- Parexel International GmbH, Early Phase Clinical Unit Berlin, Berlin, Germany

REFERENCES:
- [Derived] Ahn SS, Lee M, Baek Y, Lee S. A Randomized Pharmacokinetic Study in Healthy Male Subjects Comparing a High-concentration, Citrate-free SB5 Formulation (40 mg/0.4 ml) and Prior SB5 (Adalimumab Biosimilar). Rheumatol Ther. 2022 Aug;9(4):1157-1169. doi: 10.1007/s40744-022-00471-8. Epub 2022 Jul 1. PMID 35776269